CLINICAL TRIAL: NCT02168192
Title: Breaking Bad News in Obstetrics: A Trial of Simulation-Debrief Based Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 10-08-275
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Breaking Bad News Skills; Communications Skills; Medical Education; Obstetrics; Simulation
Keywords: Breaking bad news skills; Communications skills; Medical education; Obstetrics; Simulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Lecture (Placebo Comparator): These subjects received a 10 minute power point lecture on BBN skills.
  Interventions: Behavioral: Traditional lecture
- Simulation-Debrief (Experimental): These subjects received a formal debrief process, reviewing their prior baseline simulation.
  Interventions: Behavioral: Simulation-Debrief

INTERVENTIONS:
Behavioral: Simulation-Debrief — Subjects underwent a formal debrief, reviewing the BBN skills exhibited in their prior simulation of an obstetrical communication skills scenario.
  Arms: Simulation-Debrief
Behavioral: Traditional lecture — Control group underwent lecture for approximately 10 minutes reviewing BBN skills.
  Arms: Traditional Lecture

SUMMARY:
The purpose of this study is to assess the utility of training in Breaking Bad News (BBN) skills. We hypothesize that given little or no formal training in breaking bad news, obstetric providers will benefit from a curriculum of teaching breaking bad news techniques, but will benefit more from a simulation teaching technique than from a lecture in breaking bad news techniques.

The investigators also hypothesize that providers who have undergone breaking bad news simulation will receive improved scores after the simulation debriefing compared to their pre-simulation scores, and their improvement with be greater than the control group.

DETAILED DESCRIPTION:
The investigators' study is part of a planned educational initiative on breaking bad news communication skills, planned for house staff in the department of Obstetrics and Gynecology. All subjects will undergo both a baseline and post-education simulation. The investigators' study intervention is a personalized review and debriefing of the simulation, as compared with a conventional lecture in order to assess the best curriculum for teaching this skill set.

The investigators' study design will be described, consent obtained and consenting house staff will be randomized to participate in a simulation-based education session/debrief or to attend lecture. Randomization will be achieved using sequential opaque envelopes containing allocation cards, designating group assignment. A physician who is not involved in the study will randomly insert allocation cards into the envelopes and group assignment will be concealed until after enrollment is complete.

Subjects will be assigned a study number. The list of subject identifiers and study numbers will be kept separate from other study data, and destroyed after all phases of the study are complete. All other study data will have identifying information deleted, and will be stored in a password protected database.

The investigators plan to have subjects assess baseline characteristics and breaking bad news skills using a self-assessment tool. Subsequently all house staff will be evaluated on their management of breaking bad news through a baseline SP scenario, with assessments by physician-teachers as well as the SPs . These SPs are non-physicians, and do not have supervisory control over the study subjects. The physician-teachers are the co-investigators on this study: Drs. Chazotte, Dayal, Landsberger, Bernstein, Goffman, and Karkowsky.

After this baseline assessment, the intervention group will debrief their baseline simulation with a physician educator. The control group will instead undergo a conventional lecture about "Breaking Bad News" techniques. Finally, both groups will undergo a second simulation, which will be assessed by SPs and physician-teachers

After this step, subjects will fill out self-assessment tools on BBN. House staff who did not undergo the conventional curriculum will then attend the lecture; similarly, those subjects who were not in the intervention group will then have the opportunity to review their simulation in a personal debriefing session.

Six months after the study, we plan to have all subjects fill out a self-assessment form to assess if any long-term change to their BBN skills has been sustained.

SPs will be formally trained in the scenario and in their responses, as well as in standardized assessment of the subjects.

ELIGIBILITY:
Inclusion Criteria:

-Montefiore Medical Center Obstetrics/Gynecology department house staff.

Exclusion Criteria:

* House staff that were unable to attend at least two sessions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
BBN skills | Immediate
  As evaluated by IRB-approved evalution

SECONDARY OUTCOMES:
Subject BBN confidence | Immediately and 6 months post-intervention
  Subject BBN confidence about their communications skills in the setting of Breaking Bad news was evaluated immediately post-intervention and 6-months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Chazotte, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States